CLINICAL TRIAL: NCT02129582
Title: Phase I Trial of Escalated Doses of Targeted Marrow Irradiation (TMI) Combined With Fludarabine and Busulfan as Conditioning Regimen for Allogeneic Hematopoietic Progenitor Cell Transplantation
Brief Title: Targeted Marrow Irradiation, Fludarabine Phosphate, and Busulfan Before Donor Progenitor Cell Transplant in Treating Patients With Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE9Z13
Record Dates: First submitted 2014-04-30; First posted 2014-05-02 (Estimated); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Acute Myeloid Leukemia; Hematologic Malignancies; Acute Lymphocytic Leukemia; Non Hodgkin Lymphoma; Hodgkin Lymphoma; Multiple Myeloma; Myelodysplastic Syndrome; Chronic Lymphocytic Leukemia; Chronic Myeloid Leukemia; Myelofibrosis; Myeloproliferative Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Hematologic Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple Myeloma; Myelodysplastic Syndromes; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Primary Myelofibrosis | interventions — fludarabine phosphate; Busulfan; Antilymphocyte Serum; thymoglobulin; Tacrolimus; Methotrexate; merphos

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (TMI, fludarabine, busulfan, allogeneic HPCT) (Experimental): CONDITIONING: Patients undergo TMI BID on days -10 to -7. Patients also receive fludarabine phosphate IV over 1 hour on days -6 to -2 and busulfan IV or PO on days -5 and -4.
  TRANSPLANT: Patients undergo allogeneic hematopoietic progenitor cell transplant on day 0.
  GVHD PROPHYLAXIS: Patients receive anti-thymocyte globulin IV on days -3 and -2, tacrolimus IV or PO beginning on day -1 for at least 6 months with taper beginning at 4 months, and methotrexate IV on days 1, 3, 6, and 11.
  Interventions: Radiation: total marrow irradiation; Drug: fludarabine phosphate; Drug: busulfan; Procedure: myeloid progenitor cell transplantation; Biological: anti-thymocyte globulin; Drug: tacrolimus; Drug: methotrexate; Other: laboratory biomarker analysis

INTERVENTIONS:
Radiation: total marrow irradiation — Undergo TMI
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Drug: busulfan — Given IV or PO
  Other Names: BSF; BU; Misulfan; Mitosan; Myeloleukon
Procedure: myeloid progenitor cell transplantation — Undergo allogeneic hematopoietic progenitor cell transplant
  Other Names: MPCT
Biological: anti-thymocyte globulin — Given IV
  Other Names: ATG; ATGAM; lymphocyte immune globulin; Thymoglobulin
Drug: tacrolimus — Given IV or PO
  Other Names: FK 506; Prograf
Drug: methotrexate — Given IV
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of targeted marrow irradiation when given with fludarabine phosphate and busulfan before donor progenitor cell transplant in treating patients with hematologic malignancies. Targeted marrow irradiation is a type of specialized radiation therapy that delivers a high dose of radiation directly to the cancer cells, which may kill more cancer cells and cause less damage to normal cells. Giving targeted marrow irradiation and chemotherapy drugs, such as fludarabine phosphate and busulfan, before a donor progenitor cell transplant may help stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's progenitor cells. When the healthy progenitor cells from a donor are infused into the patient they may help the patient's bone marrow make progenitor cells, red blood cells, white blood cells, and platelets.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose of targeted marrow irradiation given in combination with fludarabine (fludarabine phosphate) and busulfan as conditioning regimen for allogeneic hematopoietic progenitor cell transplantation.

SECONDARY OBJECTIVES:

I. To describe the toxicity profile of the conditioning regimen of targeted marrow irradiation (TMI), fludarabine and busulfan for allogeneic hematopoietic progenitor transplantation.

II. To describe the use of two techniques of delivering TMI, volumetric modulated arc therapy (VMAT) and TomoTherapy, on patient's computed tomography (CT) simulation images and describe differences in organ avoidance and target coverage, planning time, and treatment delivery time.

III. To determine the disease response status 100 days after allogeneic hematopoietic progenitor cell transplantation with the conditioning regimen of TMI, fludarabine and busulfan.

IV. To determine the rates of acute graft versus host disease after allogeneic hematopoietic progenitor cell transplantation with the conditioning regimen of TMI, fludarabine and busulfan.

OUTLINE: This is a dose-escalation study of TMI.

CONDITIONING: Patients undergo TMI twice daily (BID) on days -10 to -7. Patients also receive fludarabine phosphate intravenously (IV) over 1 hour on days -6 to -2 and busulfan IV or orally (PO) on days -5 and -4.

TRANSPLANT: Patients undergo allogeneic hematopoietic progenitor cell transplant on day 0.

GRAFT-VERSUS-HOST DISEASE (GVHD) PROPHYLAXIS: Patients receive anti-thymocyte globulin IV on days -3 and -2, tacrolimus IV or PO beginning on day -1 for at least 6 months with taper beginning at 4 months, and methotrexate IV on days 1, 3, 6, and 11.

After completion of study treatment, patients are followed up at 100 days, 6 months, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients ineligible to receive full myeloablative conditioning regimen for allogeneic hematopoietic progenitor cell transplant due to age or comorbidities
* Patients must have histologically or cytologically diagnosis of hematologic malignancies with an indication for allogeneic hematopoietic progenitor cell transplantation, who are ineligible to receive a full ablative conditioning regimen as part of their transplantation, including:

  * Acute myeloid leukemia
  * Acute lymphocytic leukemia
  * Non Hodgkin lymphoma
  * Hodgkin lymphoma
  * Multiple myeloma
  * Myelodysplastic syndrome
  * Chronic lymphocytic leukemia
  * Chronic myeloid leukemia:
  * Myeloproliferative syndromes including myelofibrosis
* Complete remission is not necessary for enrollment in this protocol
* Patients must have an allogeneic hematopoietic progenitor cell donor (HPCT), either a matched sibling, mismatched (1 allele) sibling, or a matched unrelated donor (MUD) or a mismatched (1 allele) unrelated donor

  * Previous hematopoietic progenitor cell transplantation is allowed; a minimum of 6 months should have elapsed from prior autologous hematopoietic progenitor cell transplantation and a minimum of 6 months should have elapsed since prior allogeneic hematopoietic progenitor cell transplantation; prior transplantation with conditioning regimens using total body irradiation is not allowed
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy of > 12 weeks, in the opinion of and as documented by the investigator
* Patients must have adequate hepatic, and renal function as defined below: there is no exclusion for the presence of cytopenias

  * Total bilirubin ≤ 1.5 times the institutional upper limit of normal
  * Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) ≤ 2.5 X institutional upper limit of normal
  * Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 2.5 X institutional upper limit of normal
  * Creatinine clearance (calculated by the Cockroft-Gault formula) ≥ 60 ml/min
  * Pulmonary Function Tests (FEV1, FVC, DLCO) 40%.
* Women of child-bearing potential and men must agree to use adequate contraception (double barrier method of birth control or abstinence) from the time of study entry, for the duration of study participation and for 3 months after completing treatment; should a woman become pregnant or suspect that she is pregnant while she or her partner is participating in this study, she should inform the treating physician immediately
* Subjects must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior non-hematologic treatment toxicities must be resolved to ≤ grade 1 according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0, with the exception of the following grade 2 toxicities: alopecia; dry skin; spleen disorders, hearing impairment; tinnitus; hypothyroidism; hyperthyroidism; endocrine disorders; blurred vision; cataracts; constipation; gastroesophageal reflux; fatigue; abnormal coagulation tests INR and/or aPTT; weight gain or weight loss; anorexia; glucose intolerance; hypoalbuminemia; hypokalemia; muscle weakness; dysgeusia; paresthesias; peripheral motor and/or sensory neuropathy; hot flashes; hypertension.
* Patients must not have received other investigational agents within 14 days of initiation of the conditioning regimen
* Patients with untreated brain metastases should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to fludarabine and or busulfan or other agents used in this study
* Prior allogeneic hematopoietic progenitor cell transplantation
* Prior autologous hematopoietic progenitor cell transplantation if the conditioning regimen included total body irradiation
* Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements; this exclusion criterion does not include the underlying disease for which the patient is undergoing hematopoietic progenitor cell transplantation
* Pregnant or breastfeeding women are excluded from this study; breastfeeding should be discontinued
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Patients with a history of therapy with radiation therapy are excluded
* Due to technical limitations of TMI, patients must be no taller than 1.9 m (6 feet 4 inches), and no wider from elbow to elbow in the supine position than 60 cm.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-11-05 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of targeted marrow irradiation defined as the dose level immediately below that in which greater than or equal to 2/6 subjects experience a dose limiting toxicity assessed using NCI CTCAE version 4.0 | Up to day 32

SECONDARY OUTCOMES:
Incidence of toxicities assessed using NCI CTCAE version 4.0 | Up to day 32
Patient mortality | Day 100
Organ avoidance | Up to 12 months
  Will be compared between the two techniques of delivering TMI (VMAT and TomoTherapy) using patients' CT simulation images.
Target coverage | Up to 12 months
  Will be compared between the two techniques of delivering TMI (VMAT and TomoTherapy) using patients' CT simulation images.
Planning time | Up to 12 months
  Will be compared between the two techniques of delivering TMI (VMAT and TomoTherapy) using patients' CT simulation images.
Treatment delivery time | Up to 12 months
  Will be compared between the two techniques of delivering TMI (VMAT and TomoTherapy) using patients' CT simulation images.
Disease response status, assessed by standard criteria for the presence of relapse | Day 100
Rates of acute GVHD, graded and staged according to the Blood and Marrow Transplant Clinical Trials Network Manual of Operations | Up to 100 days

CONTACTS AND LOCATIONS:
Overall Officials: Molly Gallogly, MD, PhD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States